CLINICAL TRIAL: NCT00001628
Title: The Role of Angiotensin Type I Receptor in the Regulation of Human Peripheral Vascular Function
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 970140; 97-H-0140
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-06

CONDITIONS: Atherosclerosis; Heart Failure, Congestive; Hypertension; Myocardial Infarction
Keywords: Angiotensin Receptor Antagonist; Atherosclerosis; Blood Flow; Endothelium; Endothelial Dysfunction
MeSH Terms: conditions — Atherosclerosis; Heart Failure; Hypertension; Myocardial Infarction | interventions — Angiotensin II Type 1 Receptor Blockers

INTERVENTIONS:
Drug: Angiotensin II type 1 receptor antagonists

SUMMARY:
The renin angiotensin system (RAS) plays an important physiological and pathophysiological role in the control of blood pressure and plasma volume. Inhibition of the RAS is useful in the treatment of hypertension, cardiac failure and in some patients with myocardial infarction. Several recent clinical trials with angiotensin converting enzyme inhibitors (ACEI) have shown that they also reduce the incidence of myocardial infarction, but the mechanisms underlying this anti-ischemic effect are poorly understood. ACEI reduce angiotensin II synthesis and prevent bradykinin degradation. Results from ongoing studies in the Cardiology Branch (Protocol 95-H-0099) designed to investigate the link between ACEI and the vascular endothelium indicate that ACEI improve peripheral endothelial function, an effect that is partially mediated by bradykinin. The current protocol is designed to investigate whether the beneficial effects of ACEI on peripheral endothelial function are also due to inhibition of angiotensin II. The recent development of selective angiotensin II type 1 (AT1) receptor antagonists allows us to specifically examine the effects of angiotensin II on vasomotor activity.

DETAILED DESCRIPTION:
The renin angiotensin system (RAS) plays an important physiological and pathophysiological role in the control of blood pressure and plasma volume. Inhibition of the RAS is useful in the treatment of hypertension, cardiac failure and in some patients with myocardial infarction. Several recent clinical trials with angiotensin converting enzyme inhibitors (ACEI) have shown that they also reduce the incidence of myocardial infarction, but the mechanisms underlying this anti-ischemic effect are poorly understood. ACEI reduce angiotensin II synthesis and prevent bradykinin degradation. Results from ongoing studies in the Cardiology Branch (Protocol 95-H-0099) designed to investigate the link between ACEI and the vascular endothelium indicate that ACEI improve peripheral endothelial function, an effect that is partially mediated by bradykinin. The current protocol is designed to investigate whether the beneficial effects of ACEI on peripheral endothelial function are also due to inhibition of angiotensin II. The recent development of selective angiotensin II type 1 (AT1) receptor antagonists allows us to specifically examine the effects of angiotensin II on vasomotor activity.

ELIGIBILITY:
Patients over 18 years with endothelial dysfunction requiring diagnostic cardiac catheterization.

Normal volunteers or patients undergoing catheterization who have normal coronary arteries without risk factors for atherosclerosis will be used as controls.

No unstable angina.

No significant left main disease (greater than 50% stenosis).

No recent myocardial infarction (less than 1 month).

No pregnancy, lactation.

No allergy to losartan.

No renal failure (creatinine greater than 2.5 mg/dl).

Ability to withdraw ACE inhibitors.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36
Dates: Start 1997-07; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ontyd J, Schrader J. Measurement of adenosine, inosine, and hypoxanthine in human plasma. J Chromatogr. 1984 May 11;307(2):404-9. doi: 10.1016/s0378-4347(00)84113-4. No abstract available. PMID 6736187
- [Background] Cockcroft JR, Sciberras DG, Goldberg MR, Ritter JM. Comparison of angiotensin-converting enzyme inhibition with angiotensin II receptor antagonism in the human forearm. J Cardiovasc Pharmacol. 1993 Oct;22(4):579-84. doi: 10.1097/00005344-199310000-00011. PMID 7505360
- [Background] Gottlieb SS, Dickstein K, Fleck E, Kostis J, Levine TB, LeJemtel T, DeKock M. Hemodynamic and neurohormonal effects of the angiotensin II antagonist losartan in patients with congestive heart failure. Circulation. 1993 Oct;88(4 Pt 1):1602-9. doi: 10.1161/01.cir.88.4.1602. PMID 8403307